CLINICAL TRIAL: NCT05610306
Title: Quality of Life in Middle-aged and Older Patients With Congenital Ichthyosis: a Qualitative Study With In-depth Interviews
Brief Title: Quality of Life in Middle-aged and Older Patients With Congenital Ichthyosis
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2020-3226A3
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-11

CONDITIONS: Congenital Ichthyosis
MeSH Terms: conditions — Ichthyosis Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inherited ichthyosis patients: Interviews
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Qualitative interviews to gain insight into the impact of ichthyosis on the biological, psychological, and social quality of life in adult and elderly patients.

SUMMARY:
The goal of this observational study is to learn about the quality of life in patients with congenital ichthyosis.

The main question it aims to answer are:

• What is the impact of ichthyosis on the biological-psychological-social quality of life in adult and elderly patients with inherited ichthyosis ?

Participants will take part in individual interviews in which the investigators will explore if and how ichthyosis impacts their quality of life. Examples of such questions are whether participants experience pain, experience struggles in their personal or professional lives, with sports activities or if participants experience a financial burden.

DETAILED DESCRIPTION:
There is limited knowledge on factors affecting the quality of life in patients with ichthyosis, especially in middle-aged and elderly patients. With this study the investigators aim to study the impact of inherited ichthyosis on the biological-psychological-social quality of life in adult and elderly patients with ichthyosis.

Secondary research questions include:

1. What is the impact of ichthyosis on the biological quality of life; by analysing physical complaints, adverse events and drug management in patients with long-term medication use of both topical and systemic treatments, and discussing the sexual health and reproductive challenges?
2. What is the impact of ichthyosis on the psychological quality of life; by examining patients' self-esteem and any clinical symptoms of body dysmorphic disorder, and mental and emotional complaints such as concerns about their future care?
3. What is the impact of ichthyosis on the social quality of life; by analysing interpersonal relationships, social support dynamics, societal costs and awareness, and career opportunities?

Furthermore the investigators aim to discover knowledge gaps in current patient management and possible areas of improvement in patient care towards health professionals.

ELIGIBILITY:
Inclusion Criteria:

* 30 years of age and older
* Clinical or genetic confirmed variant of congenital ichthyosis

Exclusion Criteria:

* <30 years of age
* ichthyosis vulgaris
* another primary chronic skin condition besides ichthyosis
* patients who are not able to read/speak Dutch

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with congenital ichthyosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment | 1 day
  Qualitative evaluation of quality of life by interviews of patients with inherited ichthyosis.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni H Gostynski, MD, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre +, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The interview protocol of the qualitative study. Supplementary Table with patient demographics.
Supporting Information: Study Protocol, Analytic Code
Time Frame: From 22-10-2024 onwards, no end date.
Access Criteria: Everyone who accesses the ClinicalTrials.gov website will be able to view the individual participant data (IPD) and supporting information associated with the study.

DOCUMENTS (2):
  • Study Protocol (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT05610306/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT05610306/SAP_001.pdf